CLINICAL TRIAL: NCT06660758
Title: Pilot Study of the Entarik System With Advanced Functionality in Health Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gravitas Medical, Inc. (Industry)
Collaborators: Theranova, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CRD-04-1934-01
Record Dates: First submitted 2024-10-24; First posted 2024-10-28 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Healthy Adults
MeSH Terms: interventions — Enteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Healthy Adults (Experimental): An Entarik feeding tube will be introduced and subjects will receive a meal administered through the feeding tube. Ultrasound and other data will be recorded before, during and after the meal is administered.
  Interventions: Device: Feeding tube (Entarik)

INTERVENTIONS:
Device: Feeding tube (Entarik) — Feeding tube placement will be verified using multiple methods in the duodenum and stomach.

SUMMARY:
In this single-site study, data will be recorded during nasogastric or orogastric placement (and post-pyloric placement) and removal of the Entarik Feeding Tube. Data will also be collected prior to, during, and following the delivery of a meal through the feeding tube.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old
2. Able to provide informed consent
3. Capable and willing to follow all study-related procedures
4. Confirmed fasted state for a minimum of 8 hours prior to study initiation

Exclusion Criteria:

1. Inability to receive a feeding tube
2. Known self-reported history of hiatal hernia, esophagitis, esophageal strictures or gastric ulcers
3. Has a basilar skull fracture
4. Self-reports pregnancy
5. Deemed unsuitable for enrollment in study by the investigator based on subjects' history or physical examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2025-12-21 (Estimated); Study Completion 2025-12-22 (Estimated)

PRIMARY OUTCOMES:
Freedom from device-related adverse events | From enrollment to end of study (1 day)
  The incidence and severity of Adverse Events (AEs) including device and procedure-related AEs and the incidence and severity of Serious Adverse Events (SAEs) will be evaluated throughout the study.
  Based on the non-invasive nature of the device and clinical experience gained to date, there are expected to be no SAEs nor Unanticipated Adverse Device Effects (UADEs) in the study. If any SAEs or UADEs occur they will be documented and reported, but there are no planned formal hypotheses associated with the evaluation of safety.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Sorrentino, MD, Principal Investigator
Locations (1):
- Gravitas Medical, Inc., Berkeley, California, United States

IPD SHARING:
Plan to Share IPD: No
This is a device development study. Subject data may be shared at a later time at the sponsor's discretion.